CLINICAL TRIAL: NCT03192579
Title: Effect of Rosuvastatin and Eicosapentaenoic Acid on Neoatherosclerosis: The LINK-IT Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, Kobe University Graduate School of Medicine, Kobe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KobeU
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease Progression
Keywords: neoatherosclerosis
MeSH Terms: interventions — Rosuvastatin Calcium; Eicosapentaenoic Acid

STUDY DESIGN:
Intervention Model Description: Consecutive patients with stent implantation who were performed coronary angiography and OCT follow-up of the coronary arteries were screened. The patients with neoatherosclerosis were randomly assigned to either 2.5-5mg/day of rosuvastatin therapy or 10mg/day(up to 20mg) of rosuvastatin and 1800mg/day of eicosapentaenoic acid therapy at a 1:1 ratio for 12 months.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard lipid lowering therapy (Experimental): Start with only rosuvastatin 2.5mg and up to 20mg/day
  Interventions: Drug: Standard dose rosuvastatin
- Intensive lipid lowering therapy (Active Comparator): Start EPA and rosuvastatin 10mg/day and up to 20mg/day
  Interventions: Drug: EPA and high dose rosuvastatin

INTERVENTIONS:
Drug: EPA and high dose rosuvastatin — After randomization, patients with intensive lipid lowering therapy start EPA (1800mg/day) and high dose rosuvastatin (10mg/day) for 12 months.
  Other Names: Rosuvastatin; Eicosapentaenoic acid
  Arms: Intensive lipid lowering therapy
Drug: Standard dose rosuvastatin — After randomization, patients with standard lipid lowering therapy start only rosuvastatin (2.5mg/day) for 12 months.
  Other Names: rosuvastatin
  Arms: Standard lipid lowering therapy

SUMMARY:
This study aim to evaluate whether intensive lipid lowering therapy may improve the clinical outcomes in coronary artery disease patients with in-stent neoatherosclerosis, in comparison with standard therapy.

DETAILED DESCRIPTION:
Eicosapentaenoic acid and statin therapy prevents cardiovascular events. However, the impact of these treatment in patients with in-stent neoatherosclerosis (NA) has not been clarified.

Drug-eluting stent (DES) use has successfully offered a significant reduction of mid-term restenosis and repeat revascularization by controlling acute-phase excessive intimal growth after stent implantation. However, several issues still exists mainly with respect to the late-phase clinical events, including late stent thrombosis and delayed restenosis after first- and second-generation DES implantation. A growing number of evidence have suggested the potential contribution of atheromatous changes within neointimal tissue, namely neoatherosclerosis (NA) on these phenomena occurring long-term after stent implantation.

Rosuvastatin is one of the most widely used statin that has an extensive evidence for reducing adverse cardiovascular event in patients with coronary artery disease. The JUPITER (Justification for the Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin ) trial demonstrated that 20mg/del of Rosuvastatin significantly reduced combined primary end point of myocardial infarction, stroke, arterial revascularization, hospitalization for unstable angina, or death from cardiovascular causes in patients with elevated CRP level. Also, the ASTEROID Trial showed that high-intensity statin therapy with rosuvastatin of 40 mg/d reduced low-density lipoprotein cholesterol (LDL-C) level to 60.8 (20.0) mg/dL (53.2% reduction) and induced significant plaque volume reduction measured by intravascular ultrasound (IVUS) (JAMA. 2006;295:1556-1565). Although the dose of lipid-lowering therapy is one of the major contributing factors to the effect of lipid-lowering therapy, it is also well known that the effect of statin therapy has ethnic variation, being less statin dose required for Asians. Indeed in Japan, relatively less intensive statin therapy has been reported to reduce serum LDL-C level on average by 70mg/dl (change from baseline: -42%) and reduced atheroma volume measured by IVUS. Using Virtual histology IVUS, Hong et al. demonstrated that 10 mg/day Rosuvastatin therapy reduced serum low-density lipoprotein cholesterol (LDL-C) on average by 83 mg/dl (change from baseline: -32%) and decreased atheroma burden in 67% of enrolled patients.

Eicosapentaenoic acid (EPA) is another lipid-lowering therapyAccording to a recent study, the addition of highly purified EPA to statin therapy provides further benefits in preventing cardiovascular events (Yokoyama M, Origasa H, Matsuzaki M et al. Effects of eicosapentaenoic acid on major coronary events in hypercholesterolaemic patients (JELIS): a randomised open-label, blinded endpoint analysis. Lancet 2007;369:1090-8.). Also, we had reported that the concomitant use of eicosapentaenoic acid (EPA) and rosuvastatin reduced serum hs-CRP level significantly and increased fibrous cap thickness in patients who were detected thin-cap fibroatheroma by OCT.

Recently, we conducted a retrospective, nonrandomized OCT study to demonstrate that higher LDL cholesterol and CRP levels were independent determinants of NA progression. Also, Therefore, we designed a prospective, randomized OCT study in Japan to assess the effect of 10 mg/day plus eicosapentaenoic acid (EPA) versus 2.5-5.0 mg/day of rosuvastatin on the extent of NA after stent implantation.

The OCT operators randomly assigned 50 patients who were detected NA on follow-up optical coherence tomography (OCT) examination to either 2.5-5mg/day of rosuvastatin therapy (standard dose group) or 10mg/day(up to 20mg/day) of rosuvastatin and 1800mg/day of eicosapentaenoic acid therapy (intensive dose group). Serial coronary angiography and OCT were performed at 12 months after baseline OCT procedure. Sample size was calculated based on the assumption that the average difference in multiplication of lipid arc and lipid length growth between the groups receiving only rosuvastatin and EPA (1800mg/day) adding on rosuvastatin is 81.5, and the SD of multiplication of lipid arc and lipid length growth distribution for either group is 102.1. With a 2-sided alpha level of 0.05 and a power of 80%, 25 patients were required in each group.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with stent implantation who were performed coronary angiography and OCT follow-up of the coronary arteries were candidate. During this period, OCT was performed for the following reasons: 1) planned follow-up coronary angiography and OCT for routine stent follow-up or due to other study protocols, regardless of symptoms; 2) evidence of myocardial ischemia such as silent myocardial ischemia, stable angina, or acute coronary syndrome; or 3) planned follow-up angiography for other stent segments. These patients were implanted bare metal stent, sirolimus-eluting stents (Cypher, Cordis, Miami Lakes, FL, USA), paclitaxel-eluting stents (Taxus, Boston Scientific, Natick, MA, USA), or everolimus-eluting stents (XIENCE V, Abbott Vascular, Santa Clara, CA, USA). The investigators assessed their OCT examination at the follow-up OCT time and patients who were detected NA on OCT findings were eligible for the presence study.

Exclusion Criteria:

* Exclusion criteria for OCT were 1) anatomically unsuitable target artery for OCT according to previously described criteria, 10 2) apparent congestive heart failure, 3) renal insufficiency with baseline creatinine level ≥2.0 mg/dL expect for under hemodialysis, or 4) lack of written informed consent from the patient.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07-26 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Lipid index change between baseline and 12 month follow-up | Baseline and 12 month follow-up
  Lipid core arc was measured by every 0.2-mm interval throughout segments with NA on OCT findings. The mean lipid core arc was calculated for each lesion. Then, the lipid index was calculated by multiplying the mean lipid core arc by the lipid core longitudinal length.

SECONDARY OUTCOMES:
Macrophage grade change between baseline and 12 month follow-up | Baseline and 12 month follow-up
  Macrophage arc were measured on OCT images with NA every 0.2-mm intervals and divided 4 groups as follows: grade 0, no mac¬rophage; grade 1, localized macrophage accumulation (<30°); grade 2, clus¬tered accumulation ≥30° and <90°; grade 3, clus¬tered accumulation ≥90° and <270°; and grade 4, clustered accumulation ≥270° and <360° . Macrophage grade was evaluated as summation of 0 to 4 grades across all cross section in NA.

CONTACTS AND LOCATIONS:
Overall Officials: Hiromasa Otake, ph.D, Study Chair — Kobe University Graduate School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided